CLINICAL TRIAL: NCT04503161
Title: The Effect of an ASC-seeded Collagen Hydrogel on Cerebrospinal Fluid Leak Rates Following Skull Base Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left institution
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-52778
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: CSF Leak
MeSH Terms: conditions — Cerebrospinal Fluid Otorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hydrogel recipient (Experimental)
  Interventions: Device: Duragen with Collagen Hydrodel and ASCs

INTERVENTIONS:
Device: Duragen with Collagen Hydrodel and ASCs — Duragen combined with collagen hydrogel and patient's stem cells

SUMMARY:
This project seeks to test whether a cell-seeded collagen hydrogel dressing can reduce CSF leak after skull base surgery. Normally, patients at risk for CSF leak are treated with a commercial collagen matrix called Duragen. In this study, our sterile, cGMP manufactured collagen hydrogel dressing will be seeded with the stromal vascular fraction (SVF) mechanically isolated from lipoaspirate taken intra-operatively. This SVF contains pro-regenerative adipose stem cells (ASCs). The ASC-seeded hydrogel will be used as a supplement to Duragen to reinforce the skull base closure. The goal is to establish safety as well as to secondarily evaluate for effectiveness in reducing CSF leak postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18
* Planned for skull base surgery
* Able to understand and willing to sign a written informed consent form

Exclusion Criteria:

* active skull base infection
* no plan for DuraGen repair by operating surgeon

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Rate of CSF leak | 6 months active participation (date of surgery + 6 months follow up via chart review)

SECONDARY OUTCOMES:
Length of hospital stay | 6 months active participation (date of surgery + 6 months follow up via chart review)
Need for reoperation | 6 months active participation (date of surgery + 6 months follow up via chart review)
Postoperative hematoma | 6 months active participation (date of surgery + 6 months follow up via chart review)
Postoperative infection | 6 months active participation (date of surgery + 6 months follow up via chart review)
Need for rehospitalization | 6 months active participation (date of surgery + 6 months follow up via chart review)
Death | 6 months active participation (date of surgery + 6 months follow up via chart review)

IPD SHARING:
Plan to Share IPD: No